CLINICAL TRIAL: NCT01646775
Title: The Effect of Perioperative Epidural Opioids on Inflammatory Cytokines and Immune Function
Brief Title: The Effect of Epidural Fentanyl on Immune Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Albert Moore, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 11-186-SDR
Record Dates: First submitted 2012-07-11; First posted 2012-07-20 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Malignancy
Keywords: opioid; malignancy; epidural
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural bupivacaine (Experimental)
  Interventions: Drug: epidural fentanyl
- Epidural bupivacaine and fentanyl (Active Comparator)
  Interventions: Drug: epidural fentanyl

INTERVENTIONS:
Drug: epidural fentanyl — withold epidural fentanyl

SUMMARY:
Background: For cancer to grow and metastasize, inflammatory and immunologic conditions in the host must be favorable. The perioperative period provides inflammatory and immunologic changes that may be pro-malignant. Anesthetic medications, including the use of opioid medication, may contribute to these changes.

Hypothesis: The investigators hypothesize that perioperative immunologic changes in patients undergoing resection of hepatic colorectal cancer recurrence, as measured by natural killer cell function and cytokine levels, will undergo less alterations in those who receive only epidural bupivacaine, as compared to those who receive epidural bupivacaine and fentanyl.

Methods: In this double blind control trial patients with no extra-hepatic evidence of cancer, undergoing a planned curative resection of hepatic recurrence of colorectal cancer, will be randomized to receive an epidural with bupivacaine and fentanyl, or bupivacaine alone. No other perioperative opioid medication will be given, and post-operative analgesia will be supplemented with acetaminophen and gabapentin. Blood samples and pain ratings using a verbal analogue scale will be obtained preoperatively, immediately and 6 hours postoperatively, and then daily until removal of the epidural catheter. Samples will be analyzed for levels of interleukin 2, 6, 8, 10, 12, 16, 17,TNF-α, TGF α and β, MCP-1, CRP, and NK cell activity. Cytokines will be measured using a suspension bead array immunoassay kit, and NK activity will be measured using flow cytometry of isolated peripheral blood mononuclear cells exposed to the K562 cell line and treated with fluorescent antibodies to intracellular markers of activation. Data will be compared between groups using t-tests, or Mann-Whitney tests as appropriate. To demonstrate a 50% smaller decrease of NK cell activity in the bupivacaine group as compared to the bupivacaine and fentanyl group the investigators will need to randomize a total of 30 patients.

ELIGIBILITY:
Inclusion Criteria:

We will consider for inclusion any adult patient undergoing a planned curative hepatic resection of a colorectal carcinoma liver recurrence.

Exclusion Criteria:

E 3. Patients Excluded Any patient unable to communicate in English or French. Any patient with evidence of extra-hepatic metastasis. Any patient with contra-indications to epidural anesthesia, or any of the medications used in the study.

Any patient with evidence of coronary artery disease or congestive heart failure, either previously or currently.

Any patient with insulin treated diabetes. Any patient with a BMI greater than 40. Any patient who has received steroids in the past 2 months. Any patient who has taken any pain medication the week before surgery. Any pregnant or breast feeding patient. Any patient with a chronic inflammatory disease, including but not limited to Lupus, rheumatoid arthritis, and inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Natural Killer cell activity. | 24 hours

SECONDARY OUTCOMES:
Visual analogue pain scores | 4days
opioid side effects | 4 days
incidence of infections | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moore, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada